CLINICAL TRIAL: NCT04879589
Title: Phase 1, Open-Label, Single-Ascending Dose, Parallel Group Study to Determine the Pharmacokinetics, Safety, and Tolerability of ATRS-2002 Administered Subcutaneously in Healthy Adult Males
Brief Title: Phase 1 Study of ATRS-2002 in Healthy Male Adults
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study abandoned, no participants enrolled
Sponsor: Syneos Health (Other)
Collaborators: Antares Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATRS-2002-20-001
Record Dates: First submitted 2021-04-26; First posted 2021-05-10 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SC ATRS-2002 (Experimental): 3 different dosages [25mg (0.13mL) , 75mg (0.4mL) and 200mg (1.05mL)] will be tested as single SC injection into the abdomen.
  Interventions: Drug: Abiraterone Acetate
- Oral Abiraterone Acetate (Active Comparator): A single dose of 1000mg of commercially available oral formulation of abiraterone acetate will be administered to enrolled participants in Cohort 4
  Interventions: Drug: Abiraterone Acetate

INTERVENTIONS:
Drug: Abiraterone Acetate — ATRS-2002
  Other Names: Zytiga

SUMMARY:
To access the safety, tolerability, pharmacokinetics and pharmacodynamics of subcutaneously administered ATRA-2002 against commercially available oral formulation of abiraterone acetate in healthy male adults

DETAILED DESCRIPTION:
The study will be conducted in 4 dosing groups of 8 subjects each.

Thirty-two healthy adult men will be randomly assigned to a treatment cohort and will receive either a single Subcutaneous (SC) dose of ATRS-2002 (abiraterone acetate), or a single oral dose of the commercially available formulation of abiraterone acetate (Zytiga®). Additionally, for Cohorts 1 through 3, a single subject will be randomized as a sentinel subject to be dosed at least 24 hours prior to the rest of cohort (ROC).

Dosing in the abiraterone acetate SC cohorts will be sequential and will start with subjects in the lowest SC dosing cohort (i.e., 25 mg). Dosing will not begin in the next highest SC dose cohort until all safety data, as well as available PK (Pharmacokinetic) data and TT levels, from the previous cohort(s) have been reviewed by the safety review committee (SRC e.g., Sponsor and Investigator) and it has been deemed safe to proceed to the next highest dose.

Dosing in the oral abiraterone acetate cohort (Cohort 4) may begin at any time during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provide written informed consent for participation in the study.
2. Be a male 18 to 55 years of age, inclusive at the time of consent.
3. Have a body mass index (BMI) between 18 and 32 kg/m2, inclusive at screening.
4. Have a normal electrocardiogram (ECG) at screening.
5. Have normal results for hematology, biochemistry, liver function, lipids and urinalysis tests at screening and at Day -1, as defined by laboratory normal ranges. Subjects with results outside of the normal ranges that are considered to be not of clinical significance may be admitted to the study at the discretion of the Investigator.
6. Have a potassium level greater than or equal to 3.8 mEq/L.
7. Have a testosterone value within the normal range at screening.
8. Have vital signs within the normal range at screening, as defined by site standard ranges. Assessments for vital signs may be repeated up to 3 times, at the discretion of the Investigator.
9. Subjects who are not vasectomized for at least 6 months, and who are sexually active with a female partner of child bearing potential (does not include post menopausal women [absence of menses for 12 months prior to drug administration] or women who have had a hysterectomy or bilateral oophorectomy [at least 6 months prior to drug administration]) must be willing to use one of the following acceptable contraceptive methods for at least 120 days post-dose:

   1. Simultaneous use of a condom and, for the female partner, hormonal contraceptives (used since at least 4 weeks);
   2. Simultaneous use of a male condom and, for the female partner, intra-uterine contraceptive device (placed since at least 4 weeks).
10. Subjects who are not vasectomized for at least 6 months, and who are sexually active with a female partner who have had a tubal ligation from at least 6 months prior to drug administration must be willing to use a condom for at least 120 days post-dose.
11. Must be willing not to donate sperm until at least 120 days post-dose
12. Be able and willing to comply with all study procedures and agree to participate in the study program as outlined in the protocol.

Exclusion Criteria:

1. Has a known allergy to study drug or any excipients contained within the study drug.
2. Has any acute or active chronic disease. Mild conditions that only require intermittent treatment and are unlikely to interfere with study results may be permitted at the discretion of the Investigator (examples include seasonal hay fever and mild eczema).
3. Has a history of any clinically important cardiovascular, pulmonary, hepatic, renal, dermal, central nervous system (CNS), or neuromuscular disease disorders or asthma (excluding non current, childhood asthma) or diabetes or any other clinically important disorder, as determined by the Investigator.
4. Has a predisposing condition that could interfere with the absorption, distribution, metabolism, or excretion of drugs or any condition that may confound the PK analyses, particularly hepatic or renal disease, as determined by the Investigator.
5. Has a history of anaphylaxis, or other severe reaction, to a drug, food, toxin, or other exposure.
6. Has an elevated PSA level at screening.
7. Has received another investigational drug including investigational agent(s) targeting the androgen receptor within 30 days or 5 half-lives (whichever is longer) prior to the screening visit.
8. Is taking, or has taken, any prescribed or over-the-counter drug or herbal product known to modulate cytochrome P450 (CYP)17 (e.g., ketoconazole, abiraterone acetate, orteronel, galeterone, or seviteronel) in the 30 days prior to the screening visit, or is planning to take any of these medications at any time during the study.
9. Is taking, or has taken, any prescribed or over-the-counter drug, herbal, or food known to modulate CYP3A4 in the 30 days prior to the screening visit, or is planning to take any of these medications or foods at any time during the study.
10. Is taking, or has taken, any prescribed CYP2D6 substrate in the 7 days (or 5 half-lives, whichever is longer) prior to the screening visit, or is planning to take any of these medications or foods at any time during the study.
11. Has a history of alcohol abuse (regularly drinks more than 10 units of alcohol per week; 1 unit = 375 mL of beer [3.5% ABV], 100 mL of wine [13.5% ABV], or 30 mL of spirit [40% ABV]).
12. Has a positive breathalyzer test at screening or at check-in (Day -1).
13. Has a history or current evidence of abuse of licit or illicit drug substances or a positive urine drug screen for drugs of abuse at screening or before dosing. Screening of illicit drug substances include: amphetamines, methamphetamines, methadone, barbiturates, benzodiazepines, cocaine, opiates, methylenedioxymethamphetamine (MDMA), phencyclidine (PCP), and tetrahydrocannabinol (THC).
14. Currently uses tobacco-containing, e-cigarette, nicotine replacement products, or has a history of tobacco use within 3 months prior to the screening visit. Subjects must not have a lifetime history of more than the equivalent of 10 pack-years.
15. Has a positive urine cotinine test at screening or at check-in (Day -1).
16. Has donated blood or plasma within 90 days prior to the screening visit.
17. Has a history of any psychiatric conditions, which at the discretion of the Investigator will pose a risk to the subject if they were to be exposed to the IP, or which would have the potential to compromise the outcomes of the study.
18. Has a history of suicidal ideation, suicide attempts, or psychiatric hospitalizations.
19. Has a positive result for Human Immunodeficiency Virus (HIV) 1/2 antibody, hepatitis C antibody, or hepatitis B surface antigen.
20. Has a history of malignancy within the past 5 years before the screening visit, with the exception of successfully treated non-metastatic basal cell or squamous cell carcinomas of the skin.
21. Has adrenal insufficiency or has used oral or inhaled corticosteroids within the past 12 months before the screening visit. Intranasal corticosteroids may be permitted.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic assessment | Pre-dose (within 30 minutes), Post dose - 4hours, 8hours, 12hours on day 1 and then 24hours, 36hours, 48hours, 60hours, 72hours, 84hours, 96hours, 168hours, 240hours, 336hours, 504hours, 672hours
  Peak concentration (CMAX)
Pharmacodynamic assessment | Pre-dose (within 30 minutes), Post dose - 4hours, 8hours, 12hours on day 1 and then 24hours, 36hours, 48hours, 60hours, 72hours, 84hours, 96hours, 168hours, 240hours, 336hours, 504hours, 672hours
  To determine TT (total testosterone) and LH (luteinizing hormone) levels from whole blood

SECONDARY OUTCOMES:
Safety assessment | Screening (Days -28 to -2), Day -1 and Days 1,3,5 and 15
  Normal 12-Lead ECG
Safety assessment | Screening (Days -28 to -2), Predose - 4 hours, 8 hours, 12 hours, 24hours, 36hours, 48 hours, 72 hours and 96 hours. Vital signs will also be measured on Day 8, 11, 15, 22 and 29.
  Abnormal Blood pressure
Safety assessment | Screening (Days -28 to -2), Predose - 4 hours, 8 hours, 12 hours, 24hours, 36hours, 48 hours, 72 hours and 96 hours. Vital signs will also be measured on Day 8, 11, 15, 22 and 29.
  Abnormal Heart rate and respiratory rate
Safety assessment | Screening (Days -28 to -2), Predose - 4 hours, 8 hours, 12 hours, 24hours, 36hours, 48 hours, 72 hours and 96 hours. Vital signs will also be measured on Day 8, 11, 15, 22 and 29.
  Abnormal Tympanic temperature
Safety assessment | Screening (Days -28 to -2), Day -1, Day 3, Day 8, Day15 and Day 29
  Abnormal Lab tests-Hematology (Hemoglobin, hematocrit, platelets, red blood cells, white blood cells and differential)
Safety assessment | Screening (Days -28 to -2), Day -1 and Days 3, 5, 8, 11, 15, 22, and Day 29
  Abnormal Lab tests-Serum Chemistry (Urea, glucose, creatinine, sodium, potassium, chloride, bicarbonate, total protein, albumin, AST, ALT, alkaline phosphatase, total bilirubin, direct bilirubin, AM cortisol, lipid profile (screening only))
Safety assessment | Screening (Days -28 to -2) and Day 29
  Abnormal Lab tests-PSA (Prostate specific antigen)
Safety assessment | Screening (Days -28 to -2), Day -1, Day 3, Day 5, Day 15, Day 29
  Abnormal Lab tests-Urinalysis (Color, clarity/turbidity, pH, specific gravity, glucose, ketones, nitrite, leukocyte esterase, microscopy)
Local tolerability | Pre-dose, post dose-4 hours, 8hours, 12hours, 24hours, 36hours, 48hours, 72hours and 96 hours. Inspection will also be done at FU visits on Day 8, 11,15, 22 and 29
  Inspection of injection site for local reactions including erythema, edema, blistering, peeling skin, and rash)
Local tolerability | Immediately after SC dosing on day 1, 4, 8, 12, 24, 36, 48, 60, 72 and 96 hrs post dose. On day 8-to measure pain 11-point numeric pain rating scale will be used
  Pain intensity (11-point numeric pain rating scale (NPRS: 0-10) where 0=no pain and 10=the worst pain imaginable)

IPD SHARING:
Plan to Share IPD: No